CLINICAL TRIAL: NCT00433355
Title: Studies on Epstein-Barr Virus as a Possible Etiological Agent for Chronic Fatigue Syndrome
Brief Title: Epstein-Barr Virus as a Possible Cause for Chronic Fatigue Syndrome
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Gailen D. Marshall, MD, PhD, The University of Mississippi Medical Center
Other Study IDs: 2006-0265
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Chronic Fatigue Syndrome; Epstein-Barr Virus
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to understand what causes a continuing fatigue for a long time with a number of symptoms occurring at the same time (Chronic Fatigue Syndrome-CFS). Epstein Barr Virus is among the group of viruses that have been associated with a continuing fatigue for a long time with a number of symptoms occurring at the same time, but the cause is still unknown.

DETAILED DESCRIPTION:
Epstein-Barr virus (EBV) is the etiological agent for heterophile positive infectious mononucleosis (IM). It is also an oncogenic herpes virus associated with African Burkitt's lymphoma (BL),nasopharyngeal carcinoma (NPC) and AIDS-associated B-cell lymphomas. EBV is also among a group of viruses that have been associated with chronic fatigue syndrome (CFS), although the etiology of CFS still remains unknown.Findings may lead to hypothesize that EBV enzymes, such as the dUTPase, have the capacity to induce immune dysregulation of the T-cell and NK cell responses and that this immune dysregulation produces immunopathology that results in the symptoms that we call CFS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults for controls.
* Adults with chronic fatigue syndrome.

Exclusion Criteria:

* Individuals with significant medical illness in reference to immunosuppressant drug.

Note: We recruit participants in the Mississippi area who could come in our site to provide blood draw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18 y/o and above with history of CFS matched those without as to age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gailen D Marshall, M.D., PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States